CLINICAL TRIAL: NCT00493714
Title: The Impact of Acute Delirium On the Level of Distress In Patients With Advanced Cancer and Their Caregivers
Brief Title: Delirium Recall in Advanced Cancer Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0341
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Cancer; Delirium
Keywords: Advanced Cancer; Delirium; Restlessness; Confusion; Caregivers; Questionnaire
MeSH Terms: conditions — Delirium; Psychomotor Agitation; Confusion | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm 1 (Patient): Cancer patient who recently experienced confusion or restlessness.
  Interventions: Behavioral: Questionnaire
- Arm 2 (Caregiver): Caregivers of cancer patients who recently experienced confusion or restlessness.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Surveys lasting 30 minutes or more.

SUMMARY:
Primary Objectives:

1. To determine the proportion of patients who experience partial or complete recollection of symptoms of delirium and the level of distress associated with this recall.
2. To determine caregiver's level of distress associated with the patient's episode of delirium.

DETAILED DESCRIPTION:
Informed Consent for Patients:

Delirium is often seen in patients with advanced cancer. Delirium is defined as confusion and restlessness. In this study, cancer patients will be asked about their memory of experiencing delirium and the distress related to those memories. Caregivers of those patients will also be asked to participate, and they will be asked questions about their experience during these situations.

You will be tested using the Memorial Delirium Assessment Scale to see if you have recovered from your delirium. If you are still eligible to take part in this study, and both you and your caregiver agree to participate in this study; you will be asked by the research nurse to complete several questionnaires that ask questions about your mental state, any memory of experiencing delirium, the severity of the delirium, symptoms you experienced during the delirium episode, and your level of emotional distress related to that event. If you and your caregiver are asked to participate in this study; you will also be asked "open-ended" questions (questions with no wrong answers) regarding the experience you had during the severe episode of delirium; your memories of the experience, and the overall distress related to it. This conversation will be tape recorded, and it will be written down word-for-word, for the purpose of analysis. The conversation is expected to last no more than 30 minutes.

The assessments and questionnaires will be conducted only at the time of interview. No further assessments or questions will be done after the completion of the study. All information collected for the study will be kept confidential. You will be assigned a study participant number when you enroll on the study, and this number will be used (instead of your name) on all data collections, to protect your confidentiality.

This is an investigational study. Up to 100 patients and 100 caregivers will take part in this study. All will be enrolled at M. D. Anderson.

Informed Consent for Caregivers:

Delirium is often seen in patients with advanced cancer. Delirium is defined as confusion and restlessness.

In this study, you will be asked about your memory of your family member's experience of delirium, and the distress related to those memories. The patient you are caring for will also be asked to participate, and they will be asked questions about their experience during these situations.

If you are eligible to take part in this study, and both you and your family member agree to participate in this study, you will be asked by the research nurse to complete several questionnaires that ask questions about your family member's mental state, your memory of your family member's experience of delirium, the severity of the delirium, symptoms your family member experienced during the delirium episode, and your level of emotional distress related to that event. If you and your caregiver are asked to participate in this study; you will also be asked "open-ended" questions (questions with no wrong answers) regarding the experience you had during your family member's severe episode of delirium, your memories of the experience, and the overall distress related to it. This conversation will be recorded using a tape recorder, and it will be written down word for word, for the purpose of analysis. The conversation is expected to last no more than 30 minutes.

The assessments and questionnaires will be conducted only at the time of interview. No further assessments or questions will be done after the completion of the study. All information collected for the study will be kept confidential. You will be assigned a study participant number when you enroll on the study, and this number will be used (instead of your name) on all data collections, to protect your confidentiality.

This is an investigational study. Up to 100 cancer patients and 100 caregivers will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of advanced cancer, defined as local recurrent and/or metastatic.
2. History of an episode of delirium during the patient's current inpatient admission, diagnosis of delirium will be made by one of the palliative care specialists according to DSM-IV-TR criteria.
3. If the patient has a complete recovery from the episode of delirium, the patient must be approached within 3 days for the possibility of inclusion in study. "Complete recovery" will be defined as diagnosis of complete resolution of all symptoms of delirium according to DSM-IV-TR criteria by one of the palliative care specialists.
4. Ability to communicate in the English language.
5. Caregiver who is 18 years of age or older (assessments used in this study have not been validated in pediatric population), is able to communicate in English and comprehend the assessment questionnaire, and is at the bedside for a significant length of time (approximately 4 hours) each day during the delirium episode. Both the patient and their caregiver must agree to participate for inclusion in the study.
6. Written informed consent signed by the patients and the participating caregivers.
7. MDAS [Memorial Delirium Assessment Scale] < 13 (Scores of 13 or above likely reflect the presence of delirium).
8. Patients will be recruited from the palliative care mobile team or the inpatient palliative care unit.

Exclusion Criteria:

1. Refusal of both the patient and their caregiver to complete assessments
2. Inability to complete assessment due to sensorial deficits other than cognition; e.g. blindness, deafness, aphasia, etc., that might impact the patient's ability to recall the episode of delirium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Advanced cancer patient having had an episode of delirium with complete recover; and their caregivers, age 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2005-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Patient Level of Distress as related to Level of Delirium | 2 Years
  Level of distress patients experience associated with delirium recall, made on a 0-4 numerical rating scale with 0=not at all and 4=extremely distressed. Summarized as a median score and as the most frequent response.
Number of patients who have partial or complete memory of experiencing any signs of delirium (confusion or restlessness) | 2 Years
  Interview with full assessment including demographic information, MMSE (Mini-Mental State Exam), DEQ (The Delirium Experience Questionnaire), and Delirium Recall Questionnaire for patient who experience complete recovery from an episode of delirium

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org